CLINICAL TRIAL: NCT00000827
Title: A Phase I/II Study of Hyperimmune IVIG in Slowing Progression of Disease in HIV-Infected Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: North American Biologicals Inc (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 273; 11249 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Immunoglobulins, Intravenous; Immunization, Passive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex

INTERVENTIONS:
Drug: Anti-HIV Immune Serum Globulin (Human)

SUMMARY:
To evaluate the safety, tolerance, pharmacokinetics, and antiviral activity of human anti-HIV immune serum globulin ( HIVIG ) at three dosage levels in HIV-infected children.

Passive antibody therapy has been used with limited success in treating advanced HIV disease in adults. HIVIG is manufactured from HIV antibody-rich plasma taken from asymptomatic donors. It is hypothesized that HIVIG will decrease the viral burden of moderately advanced HIV-positive children.

DETAILED DESCRIPTION:
Passive antibody therapy has been used with limited success in treating advanced HIV disease in adults. HIVIG is manufactured from HIV antibody-rich plasma taken from asymptomatic donors. It is hypothesized that HIVIG will decrease the viral burden of moderately advanced HIV-positive children.

Children are randomized to receive HIVIG every 4 weeks for 6 months at one of three dose levels, then are followed for 3 months after the final infusion.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* PCP prophylaxis according to CDC guidelines.

Allowed:

* Varicella-zoster immunoglobulin.
* Hepatitis B immunoglobulin.
* Prophylactic therapies not involving immunoglobulin.

Patients must have:

* HIV infection.
* CD4 count > 200 cells/mm3 (ages 2-5 years) or > 100 cells/mm3 (age > 5 years).
* Antiretroviral therapy for at least 6 months, with no change in regimen for at least 3 months prior to study entry.
* Plasma ICD p24 >= 70 pg/ml that is stable or increasing prior to study entry.
* Life expectancy of at least 6 months.

Prior Medication: Required:

* Antiretroviral therapy for at least 6 months, with stable dose for at least 3 months.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Severe diarrhea, nephrotic syndrome, or other protein-losing state that requires large doses of IVIG.
* Any other condition requiring dosing with IVIG (e.g., ITP, hypogammaglobulinemia).
* Acute illness with temperature >= 100 F and/or with IV antibiotics.
* Grade 3 or worse clinical toxicities.
* Unable to tolerate IV infusions at a minimum rate of 0.02 ml/kg/min.
* Concomitant participation in an experimental antiretroviral or HIV vaccine trial.

Concurrent Medication:

Excluded:

* IVIG.
* Chemotherapy for an active malignancy.
* MMR or rubella vaccinations.
* Intramuscular immunoglobulin.

Patients with the following prior condition are excluded:

* History of severe reaction to IVIG.

Prior Medication:

Excluded:

* IVIG within the past 60 days.
* Chemotherapy for an active malignancy within the past year.
* MMR or rubella vaccinations within the past 6 months.
* Intramuscular immunoglobulin within the past 60 days.

Ongoing drug or alcohol abuse.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45
Dates: Study Completion 1998-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stiehm ER, Study Chair; Wara DW, Study Chair
Locations (39):
- United States (37):
  - UAB, Dept. of Ped., Div. of Infectious Diseases, Birmingham, Alabama
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - Usc La Nichd Crs, Los Angeles, California
  - Childrens Hosp. LA - Dept. of Ped., Div. of Clinical Immunology & Allergy, Los Angeles, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - Children's Hosp. & Research Ctr. Oakland, Ped. Clinical Research Ctr. & Research Lab., Oakland, California
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Univ. of Connecticut Health Ctr., Dept. of Ped., Farmington, Connecticut
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Children's National Med. Ctr., ACTU, Washington D.C., District of Columbia
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - Emory Univ. School of Medicine, Dept. of Peds., Div. of Infectious Diseases, Atlanta, Georgia
  - Univ. of Maryland Med. Ctr., Div. of Ped. Immunology & Rheumatology, Baltimore, Maryland
  - Johns Hopkins Hosp. & Health System - Dept. of Peds., Div. of Infectious Diseases, Baltimore, Maryland
  - BMC, Div. of Ped Infectious Diseases, Boston, Massachusetts
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - Baystate Health, Baystate Med. Ctr., Springfield, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Children's Hospital of Michigan NICHD CRS, Detroit, Michigan
  - St. Joseph's Hosp. & Med. Ctr. of New Jersey, Paterson, New Jersey
  - Children's Hospital at Albany Medical Center, Dept. of Peds., Albany, New York
  - SUNY Downstate Med. Ctr., Children's Hosp. at Downstate NICHD CRS, Brooklyn, New York
  - North Shore-Long Island Jewish Health System, Dept. of Peds., Great Neck, New York
  - Columbia IMPAACT CRS, New York, New York
  - Incarnation Children's Ctr., New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - NYU Med. Ctr., Dept. of Medicine, New York, New York
  - Strong Memorial Hospital Rochester NY NICHD CRS, Rochester, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania
  - Med. Univ. of South Carolina, Div. of Ped. Infectious Diseases, Charleston, South Carolina
  - St. Jude/UTHSC CRS, Memphis, Tennessee
  - Children's Med. Ctr. Dallas, Dallas, Texas
  - Texas Children's Hosp. CRS, Houston, Texas
  - UW School of Medicine - CHRMC, Seattle, Washington
- Puerto Rico (2):
  - San Juan City Hosp. PR NICHD CRS, San Juan
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan

REFERENCES:
- [Background] Stiehm ER, Fletcher CV, Mofenson LM, Palumbo PE, Kang M, Fenton T, Sapan CV, Meyer WA, Shearer WT, Hawkins E, Fowler MG, Bouquin P, Purdue L, Sloand EM, Nemo GJ, Wara D, Bryson YJ, Starr SE, Petru A, Burchett S. Use of human immunodeficiency virus (HIV) human hyperimmune immunoglobulin in HIV type 1-infected children (Pediatric AIDS clinical trials group protocol 273). J Infect Dis. 2000 Feb;181(2):548-54. doi: 10.1086/315224. PMID 10669338